CLINICAL TRIAL: NCT07130682
Title: 2-fraction Stereotactic Body Proton Therapy (SBPT) With Magnetic Resonance Imaging (MRI) Guidance in Localized Prostate Cancer: A Single-arm Phase II Non-randomized Trial
Brief Title: Two-fraction Proton Therapy With MRI Guidance for Prostate Cancer: A Phase II Trial
Acronym: PT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC-2025-08
Record Dates: First submitted 2025-07-28; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer Patients Treated by Radiotherapy
Keywords: Proton Therapy; Clinician reported outcome; patient reported outcome; low or intermediate risk prostate cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 2-fraction Proton therapy (Experimental)
  Interventions: Radiation: Pencil Beam Proton Therapy Treatment Machine

INTERVENTIONS:
Radiation: Pencil Beam Proton Therapy Treatment Machine — 2 fractions will be delivered to treat low- or intermediate- risk prostate cancer

SUMMARY:
This study is testing a shorter treatment method for prostate cancer using proton therapy (PT), which is very precise and may cause fewer side effects compared to traditional radiation. However, it is expensive and not easily accessible for many patients. To make it more affordable and accessible, this study is testing whether 2 fractions of stereotactic body proton therapy (SBPT) can be as safe and effective as the standard 5 sessions.

DETAILED DESCRIPTION:
Proton therapy is an advanced form of radiation that precisely targets tumors while minimizing damage to healthy tissues. However, its high cost has limited patient access. For prostate cancer, studies have already shown that ultra-short radiation courses (as few as 2-5 sessions) using conventional X-ray-based stereotactic body radiation therapy (SBRT) provide excellent results with manageable side effects. This study aims to investigate whether 2-fraction stereotactic body proton therapy (SBPT) with magnetic resonance imaging (MRI) guidance and real-time on-board tumor tracking can achieve similar safety and efficiency as the standard 5-fraction SBPT, with the added benefit of lower costs and greater convenience for patients.

ELIGIBILITY:
Inclusion Criteria:

* Men aged < 18 years with histologically confirmed low- or intermediate-risk prostate cancer per NCCN guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* Ability to undergo magnetic resonance imaging (MRI) simulation scans without absolute contraindications, such as cardiac implantable electronic devices
* Ability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire

Exclusion Criteria:

* History of inflammatory bowel disease or other cancers (except prostate cancer)
* Prior pelvic radiotherapy, chemotherapy, radical prostatectomy, cryosurgery, or focal therapy (e.g. high-intensity focused ultrasound [HIFU]) for prostate cancer
* History of bladder neck or urethral stricture
* Transurethral resection of the prostate (TURP) < 8 weeks prior to SBPT
* Prostate volume > 100cc on MRI
* Unilateral or bilateral hip replacements
* Nodal or distant metastases, as indicated by computed tomography (CT), MRI, or prostate-specific membrane antigen (PSMA) positron emission tomography (PET) scans
* Previous androgen deprivation therapy (ADT) lasting more than 6 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study focused on the prostate cancer, which only occur in male.
Enrollment: 35 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2033-01-02 (Estimated); Study Completion 2033-06-02 (Estimated)

PRIMARY OUTCOMES:
Clinician-reported grade 2 or above genitourinary and gastrointestinal toxicity | 3 months and 24 months after treatment completion with a minimum of 24 months of follow-up and an average of 5 years.
  Genitourinary and gastrointestinal toxicity were evaluated based on the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) developed by the National Cancer Institute (NCI). Adverse effects within 3 months post-treatment are classified as acute toxicities, while those occurring after 3 months are considered late toxicities.

SECONDARY OUTCOMES:
Change in patient reported gastrointestinal and genitourinary symptoms | before treatment to 3-months and 24-months after treatment completed
  Gastrointestinal and genitourinary health-related quality of life (HQOL) are measured using the Expanded Prostate Cancer Index Composite (EPIC) questionnaire, which is a validated comprehensive instrument to measure the health-related quality of life among men with prostate cancer. EPIC consists of 5 primary domains, including urinary function, bowel habits, sexual function, hormonal functions, and overall satisfaction. Responses to each question form a Likert scale and are transformed to a 0-100 scale for each domain and subdomain, higher scores representing better HQOL.
Biochemical Progression Free Survival (bPFS) | Treatment completion date to 5 years follow-up
  Biochemical progression-free survival (bPFS) among participants will be assessed during clinical follow-up. bPFS is defined as the duration of time a localized prostate cancer patient remains free from biochemical recurrence after treatment. Biochemical recurrence is defined as a prostate-specific antigen (PSA) increase of 2 ng/mL above the nadir based on the Phoenix criteria (nadir + 2 ng/mL), confirmed by a second PSA value obtained three or more weeks later.
Distant Metastasis Free Survival | Treatment completion date to 5 years follow-up
  Distant metastasis (DM) refers to the spread of cancer cells from the prostate to distant sites outside the pelvic region. DF will be assessed during clinical follow-up using prostate-specific membrane antigen positron emission tomography (PSMA-PET), MRI, and/or other clinical imaging in cases of persistent PSA progression or emergence of symptoms. Distant metastasis free survival is defined as the duration of time from treatment completion date to the date of distant metastasis diagnosis by clinical imaging or death.
Local Failure-Free Survival (LFFS) | Treatment completion date to 5 years follow-up
  Local Failure (LF) refers to recurrent prostatic mass diagnosed by digital rectal examination, clinical imaging techniques like PSMA-PET and/or MRI, or histopathological confirmation of recurrence by biopsy. Local failure-free survival is defined as the duration of time from treatment completion date to date of local failure diagnosis or death.
Regional Failure Free Survival (RFFS) | Treatment completion date to 5 years follow-up
  Regional Failure (RF) refers to recurrent in the regional lymph nodes diagnosed by clinical imaging techniques like PSMA-PET and/or MRI. Regional failure-free survival is defined as the duration of time from treatment completion date to date of regional failure diagnosis or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Sanatorium and Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The IPD cannot be shared due to hospital policy, which restricts the sharing of patient data-even in de-identified or masked form-to ensure compliance with privacy regulations and ethical safeguards.

REFERENCES:
- [Background] Kishan AU, Ma TM, Lamb JM, Casado M, Wilhalme H, Low DA, Sheng K, Sharma S, Nickols NG, Pham J, Yang Y, Gao Y, Neylon J, Basehart V, Cao M, Steinberg ML. Magnetic Resonance Imaging-Guided vs Computed Tomography-Guided Stereotactic Body Radiotherapy for Prostate Cancer: The MIRAGE Randomized Clinical Trial. JAMA Oncol. 2023 Mar 1;9(3):365-373. doi: 10.1001/jamaoncol.2022.6558. PMID 36633877
- [Background] Westley RL, Biscombe K, Dunlop A, Mitchell A, Oelfke U, Nill S, Murray J, Pathmanathan A, Hafeez S, Parker C, Ratnakumaran R, Alexander S, Herbert T, Hall E, Tree AC. Interim Toxicity Analysis From the Randomized HERMES Trial of 2- and 5-Fraction Magnetic Resonance Imaging-Guided Adaptive Prostate Radiation Therapy. Int J Radiat Oncol Biol Phys. 2024 Mar 1;118(3):682-687. doi: 10.1016/j.ijrobp.2023.09.032. Epub 2023 Sep 29. PMID 37776979
- [Background] Wolfe S, Diven MA, Marciscano AE, Zhou XK, Kishan AU, Steinberg ML, Miccio JA, Camilleri P, Nagar H. A randomized phase II trial of MR-guided prostate stereotactic body radiotherapy administered in 5 or 2 fractions for localized prostate cancer (FORT). BMC Cancer. 2023 Sep 30;23(1):923. doi: 10.1186/s12885-023-11430-z. PMID 37777738
- [Background] Fredman E, Moore A, Icht O, Tschernichovsky R, Shemesh D, Bragilovski D, Kindler J, Golan S, Shochet T, Limon D. Acute Toxicity and Early Prostate Specific Antigen Response After Two-Fraction Stereotactic Radiation Therapy for Localized Prostate Cancer Using Peri-Rectal Spacing-Initial Report of the SABR-Dual Trial. Int J Radiat Oncol Biol Phys. 2024 Dec 1;120(5):1404-1409. doi: 10.1016/j.ijrobp.2024.06.038. Epub 2024 Jul 11. PMID 39002849
- [Background] Widmark A, Gunnlaugsson A, Beckman L, Thellenberg-Karlsson C, Hoyer M, Lagerlund M, Kindblom J, Ginman C, Johansson B, Bjornlinger K, Seke M, Agrup M, Fransson P, Tavelin B, Norman D, Zackrisson B, Anderson H, Kjellen E, Franzen L, Nilsson P. Ultra-hypofractionated versus conventionally fractionated radiotherapy for prostate cancer: 5-year outcomes of the HYPO-RT-PC randomised, non-inferiority, phase 3 trial. Lancet. 2019 Aug 3;394(10196):385-395. doi: 10.1016/S0140-6736(19)31131-6. Epub 2019 Jun 18. PMID 31227373
- [Background] Fransson P, Nilsson P, Gunnlaugsson A, Beckman L, Tavelin B, Norman D, Thellenberg-Karlsson C, Hoyer M, Lagerlund M, Kindblom J, Ginman C, Johansson B, Bjornlinger K, Seke M, Agrup M, Zackrisson B, Kjellen E, Franzen L, Widmark A. Ultra-hypofractionated versus conventionally fractionated radiotherapy for prostate cancer (HYPO-RT-PC): patient-reported quality-of-life outcomes of a randomised, controlled, non-inferiority, phase 3 trial. Lancet Oncol. 2021 Feb;22(2):235-245. doi: 10.1016/S1470-2045(20)30581-7. Epub 2021 Jan 11. PMID 33444529
- [Background] Tree AC, Ostler P, van der Voet H, Chu W, Loblaw A, Ford D, Tolan S, Jain S, Martin A, Staffurth J, Armstrong J, Camilleri P, Kancherla K, Frew J, Chan A, Dayes IS, Duffton A, Brand DH, Henderson D, Morrison K, Brown S, Pugh J, Burnett S, Mahmud M, Hinder V, Naismith O, Hall E, van As N; PACE Trial Investigators. Intensity-modulated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-B): 2-year toxicity results from an open-label, randomised, phase 3, non-inferiority trial. Lancet Oncol. 2022 Oct;23(10):1308-1320. doi: 10.1016/S1470-2045(22)00517-4. Epub 2022 Sep 13. PMID 36113498
- [Background] Santos A, Penfold S, Gorayski P, Le H. The Role of Hypofractionation in Proton Therapy. Cancers (Basel). 2022 May 2;14(9):2271. doi: 10.3390/cancers14092271. PMID 35565400
- [Background] Vidal M, Moignier C, Patriarca A, Sotiropoulos M, Schneider T, De Marzi L. Future technological developments in proton therapy - A predicted technological breakthrough. Cancer Radiother. 2021 Oct;25(6-7):554-564. doi: 10.1016/j.canrad.2021.06.017. Epub 2021 Jul 13. PMID 34272182
- [Background] Schippers JM, Lomax A, Garonna A, Parodi K. Can Technological Improvements Reduce the Cost of Proton Radiation Therapy? Semin Radiat Oncol. 2018 Apr;28(2):150-159. doi: 10.1016/j.semradonc.2017.11.007. PMID 29735191

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT07130682/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT07130682/ICF_001.pdf